CLINICAL TRIAL: NCT07090811
Title: Streamlined One-wire Logistics Optimize Transcatheter Aortic Valve Replacement
Acronym: SOLO-TAVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solo Pace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100288
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Replantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Fusion System (Experimental)
  Interventions: Device: Aortic valve repair/replacement

INTERVENTIONS:
Device: Aortic valve repair/replacement — TAVR or valvuloplasty using the Fusion System for delivery of the treatment system and for temporary rapid pacing

SUMMARY:
The goal of this study is to determine the safety and performance of a new guidewire and pacing system called the Fusion System in treating patients undergoing transcatheter aortic valve replacement (TAVR) or similar procedures. The main questions it aims to answer are:

Is the Fusion System safe? Is the Fusion System's clinical performance acceptable?

Participants will asked to sign a study consent and report any adverse events experienced until they are discharged from hospital (or a maximum of 2 days following their procedure).

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for a THV or BAV procedure in accordance with standard institutional protocols requiring temporary pacing.
2. Willing and able to comply with the follow-up evaluations
3. Been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

1. Undergoing an emergent procedure
2. An ST elevation myocardial infarction (STEMI) within 7 days of procedure
3. Had cardiac arrest within 7 days of procedure requiring CPR or defibrillation
4. An indication to require mechanical cardiac support (MCS) post-procedure
5. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical circulatory support within 30 days prior to index procedure
6. Active endocarditis within 30 days prior to index procedure
7. Cardiac imaging evidence of intracardiac mass, thrombus, or vegetation
8. Severe aortic annular or sub annular calcium per operator evaluation.
9. Bicuspid aortic valve stenosis WITH severe raphe calcium per operator evaluation.
10. Had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 90 days of index procedure
11. Severe peripheral vascular disease that would preclude safe placement of an introducer sheath
12. A planned alternative (i.e., non-femoral) access site
13. A comorbidity that would preclude index procedure or use of the Solo Pace Fusion System
14. A known, untreated neurological, psychological, psychiatric or other disorder that would interfere with trial endpoints or with cooperation with the requirements of the trial
15. Participating in another investigational drug or device study
16. Pregnant, lactating, or plan to become pregnant during the study (women of child-bearing potential must have a pregnancy test).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Transcatheter heart valve device migration/embolization or inability to complete BAV procedure. | Intraprocedure
  Incidence of failure of the Solo Pace Fusion System to provide adequate pacing leading to transcatheter heart valve device migration/embolization or the inability to complete the BAV procedure
Successful deployment of THV or BAV system over the Fusion Guidewire | Intraprocedure
  The Primary Performance Endpoint for the study consists of the following criteria (note: both criteria must be met):
  * Successful delivery to the intended position and successful deployment of a commercially available THV or BAV delivery system over the Fusion Guidewire
  * Successful pacing during THV or BAV deployment in unipolar configuration using the Fusion System